CLINICAL TRIAL: NCT03387930
Title: The Role of Lumbar Multifidus Characteristics in the Development of Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Oulu (Other); The University of Hong Kong (Other); Rush University (Other); Concordia University, Montreal (Other); Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20151027007
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
Keywords: Low back pain; lumbar multifidus; Proprioception; Elastography; Magnetic resonance imaging
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain group: Participants will be followed up over 2 years to monitor the course of low back pain
- Asymptomatic group: Participants will be followed up over 2 years to monitor the incidence and course of low back pain

SUMMARY:
Low back pain (LBP) is a severe epidemic in the world. Despite its high prevalence, 90% of the cases have no identifiable cause. Approximately 44% of them experience recurrent LBP within one year and 10% of them develop chronic LBP that lasts for three months or more.

Mechanically, the lumbar spine is unstable and requires spinal muscle to maintain spinal stability and to prevent injuries. Lumbar multifidus (LM) muscle is thought to be the major spinal stabilizer responsible for spinal stability and spinal proprioception. Prior studies have revealed that increased fat infiltration, atrophy or activation deficits of LM in patients with LBP as compared to asymptomatic individuals. Unfortunately, inconsistent findings have also been reported.

Although prior research attempted to determine if abnormal LM characteristics can inform clinical decision-making, their results are limited because they only investigated a single LM characteristic at a time, which might not reflect the actual LM condition. Further, many studies adopted cross-sectional design that could not reveal the casual relations between abnormal LM characteristics and LBP. As such, the current study aims to identify specific LM characteristics that can predict new episode of LBP in asymptomatic individuals, and recurrent/chronic LBP in individuals with LBP at baseline.

DETAILED DESCRIPTION:
Low back pain (LBP) is a severe epidemic in the world. Despite its high prevalence, 90% of the cases have no identifiable cause. While most people with LBP recover shortly after onset, approximately 44% of them experience recurrent LBP within one year and 10% of them develop chronic LBP that lasts for three months or more.

Mechanically, the lumbar spine is unstable and requires spinal muscle to maintain spinal stability and to prevent injuries. Lumbar multifidus (LM) muscle is thought to be the major spinal stabilizer responsible for spinal stability and spinal proprioception. Different cross-sectional studies have revealed that increased fat infiltration, atrophy or activation deficits of LM in patients with LBP as compared to asymptomatic individuals. Research has shown that abnormal morphology or activation of LM is associated with LBP intensity/location, or LBP-related disability. Unfortunately, inconsistent findings have also been reported.

Although prior research attempted to determine if abnormal LM characteristics can inform clinical decision-making, their results are limited because they only investigated a single LM characteristic at a time, which might not reflect the actual LM condition. Further, many studies adopted cross-sectional design that could not reveal the casual relations between abnormal LM characteristics and LBP.

Given the above, the current study aims to identify specific LM characteristics that can predict new episode of LBP in asymptomatic individuals, and recurrent/chronic LBP in individuals with LBP at baseline.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 65 years
* Symptomatic participants should have LBP that requires medical consultation(s) in the last three months
* LBP intensity of at least 5 on the 11-point numeric pain rating scale at baseline (for symptomatic participants)
* Asymptomatic participants should be pain free at baseline, and should not have LBP in the last year nor LBP lasting more than a week in the last 3 years

Exclusion Criteria:

* a history of neurological disease or vestibular impairment
* systemic inflammatory disease
* prior spinal surgery
* acute/chronic neuropathy or radiculopathy
* spinal infections/fractures/tumors, metabolic disorders,
* medical 'red flags'

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic participants should have LBP that requires medical consultation(s) in the last three months, and have LBP intensity of at least 5 on the 11-point numeric pain rating scale at baseline.
  Asymptomatic participants should be pain free at baseline, and should not have LBP in the last year nor LBP lasting more than a week in the last 3 years.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
11-point numeric pain rating scale (NPRS) for low back pain | 2 years
  The current pain intensity of each participant will be quantified by an 11-point NPRS, where 0 means no pain and 10 means the worst imaginable pain.

SECONDARY OUTCOMES:
Morphometry of lumbar multifidus | 2 years
  B-mode ultrasound imaging will be used to quantify morphometry of multifidus
Proprioception of lumbar multifidus | 2 years
  An established protocol to measure proprioception of lumbar multifidus
Stiffness of lumbar multifidus | 2 years
  Elastography will be used to measure lumbar multifidus stiffness
Fatty infiltration of lumbar multifidus | 2 years
  Magnetic resonance imaging will be used to quantify the fatty infiltration of multifidus

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No